CLINICAL TRIAL: NCT05948618
Title: Improving PRO Interpretation At the Individual Level for Patients with Cancer Using Conversational Agents and Data Visualization - Aim 3
Brief Title: Improving PRO for Patients with Cancer Using ECAs and Data Visualization
Acronym: ECA-PRO Aim 3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H-44542
Record Dates: First submitted 2023-05-19; First posted 2023-07-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: cancer; patient reported outcomes; medication adherence
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The team statistician will be blinded to experimental condition to reduce the possibility of bias. Only after analyses have been completed will the blinds be revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Embodied Conversational Agent (Experimental): The ECA systems compromises 1) a smartphone based ECA patient interface; 2) clinician authoring tool, to enable new measurement systems to be rapidly configured 3) clinician and patient data visualizations; and 4) a central server with relation database, administrative user interfaces and ability to send asynchronous notifications to users' smartphones.
  Interventions: Behavioral: Embodied Conversational Agent
- RedCap Survey (Active Comparator): An internet-based measure will use PROMIS Profile measures which will include depression, anxiety, fatigue, pain intensity and interference, sleep disturbance, physical function and satisfaction with social role
  Interventions: Behavioral: REDCap Survey

INTERVENTIONS:
Behavioral: Embodied Conversational Agent — The ECA- PRO measures will included PROMIS Profile measures, which include depression, anxiety, fatigue, pain intensity, and interference, fatigue, sleep disturbance, physical function, and satisfaction with social roles. In order to reduce boredom and confusion, equivalent forms of different items will be selected from the items pools. In this way, participants are not answering the same questions twice within one session.
  Arms: Embodied Conversational Agent
Behavioral: REDCap Survey — An internet-based measure will use PROMIS Profile measures which will include depression, anxiety, fatigue, pain intensity and interference, sleep disturbance, physical function and satisfaction with social role
  Arms: RedCap Survey

SUMMARY:
Over the past decade, the investigators have developed and tested a toll with the potential to enhance PROs at the individual level- embodied conversational agents (ECA), which are computer characters that simulate face-to-face conversation using voice, hand gestures, gaze cues, and other nonverbal behavior. The investigators have successfully used ECAs in behavioral interventions for populations with limited health literacy, elderly patients, and patients with cancer. Face-to-face encounters, in conjunction with written instructions supported by pictures, remains one of the best methods for communicating information in general but is particularly effective for individuals with limited health literacy. The investigators have also demonstrated that ECAs can be used as valid alternatives to standard paper-based surveys for substance use screening, and that the display of empathy for patients and other relational behavior by ECAs leads to increased engagement by patients over time.

DETAILED DESCRIPTION:
There is increasing recognition of the important of patient-reported outcomes (PROs) for assessment of health-related quality of life in both research and clinical settings. PROs are especially important for inherently subjective but crucial clinical phenomena such as pain, mood, and fatigue. PROs can also provide valid assessments of health where performance-based objective measures are possible, but cost prohibitive or complicated. Despite much research on PROs, concerns about reliability and validity persist, especially when used at the individual level, particularly among patients who may struggle to understand PRO questions, such as those with low health literacy.

Over the past decade, the investigators have developed and tested a tool with the potential to enhance PROs at the individual level - embodied conversational agents (ECA), which are computer characters that simulate face-to-face conversation using voice, hand gestures, gaze cues and other nonverbal behavior. The investigators have successfully used ECAs in behavioral interventions for populations with limited health literacy, elderly patients, and patients with cancer. Face-to-face encounters, in conjunction with written instructions supported by pictures, remains one of the best methods for communicating information in general, but is particularly effective for individuals with limited health literacy. The investigators have also demonstrated that ECAs can be used as valid alternatives to standard paper-based surveys for substance use screening, and that the display of empathy for patients and other relational behavior by ECAs leads to increased engagement by patients over time.

The goal of this study is to adapt our prior work on ECAs to produce ECA-PRO, a framework for administering PROs over time using an ECA. ECA-PRO will be used to administer PROs from the Patient-Reported Outcomes Measurement Information System (PROMIS), as well as measures from the Common Terminology Criteria for Adverse Events (CTCAE). The plan is to administer PROMIS measures relevant to cancer including physical functioning, fatigue, depression, anxiety, and pain interference. This study will test the system in an RCT with 100 patients receiving chemotherapy and/or radiation therapy for gastrointestinal or head and neck cancer. Participants will be randomized to provide data for 6 weeks using ECA-PRO (n=50) versus standard web administration (REDCap) (n=50).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or older
* Able to read and speak english
* Can independently consent
* Must have adequate corrected vision to use the ECA system (based on a 1 minute ECA functional screener)
* Must have adequate hearing to use the ECA system.
* Has a diagnosis of gastrointestinal cancer or head and neck cancer for which they are currently receiving chemotherapy and/or radiation treatment.
* Provider subjects must be practicing oncologists at BMC.

Exclusion Criteria:

* If the subject is incarcerated
* If the subject plans to leave the Boston area in the next 6 weeks
* Is not able to use the ECA screener

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The degree of missing data will be investigated to gauge the extent to which patients are actively engaging with the ECA-PRO system. | 6 weeks
  Assessing the completeness of the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) survey questions, taking into account the number of items that have been satisfactorily completed. By examining prevalence of missing data, the investigators aim to infer the level of patient utilization of the ECA-PRO system.

SECONDARY OUTCOMES:
Physical function | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of their symptoms related to their physical functioning. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).
Fatigue | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of their symptoms related to fatigue. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).
Depression | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of their depression symptoms. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).
Anxiety | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of their anxiety symptoms. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).
Pain Interference | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of pain interference. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).
Sleep Disturbance | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of their sleep disturbance. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).
Ability to participate in social roles and activities | 6 weeks
  There will be items from the PRO-CTCAE survey questions, that will ask participants to report the frequency of their pain and how it impacts their ability to participate in social roles and activities. Participants will fill out this survey with the ECA or in REDCap (depending on the intervention participants are receiving).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No